CLINICAL TRIAL: NCT02425826
Title: A Phase 4, Multicenter, Randomized, Placebo-controlled, Double-blind, Study of the Efficacy and Safety of Apremilast (CC-10004) in Subjects With Moderate Plaque Psoriasis
Brief Title: A Phase 4 Study of Efficacy and Safety of Apremilast in Subjects With Moderate Plaque Psoriasis.
Acronym: UNVEIL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CC-10004-PSOR-012; NCT02555826 (obsolete NCT alias)
Expanded Access: NCT03740516 (No longer available)
Record Dates: First submitted 2015-04-03; First posted 2015-04-24 (Estimated); Results first posted 2017-06-06 (Actual); Last update posted 2023-06-05 (Actual); Status verified 2020-04

CONDITIONS: Parapsoriasis
Keywords: Parapsoriasis; Plaque Psoriasis; CC-10004; Apremilast; Moderate Plaque Psoriasis; Safety
MeSH Terms: conditions — Parapsoriasis | interventions — apremilast

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Apremilast (Experimental): Apremilast 30 mg tablets orally twice daily (BID) weeks 0 to 52.
  Interventions: Drug: Apremilast; Drug: Placebo; Drug: Placebo-Apremilast
- Placebo (Placebo Comparator): Placebo tablets BID during Weeks 0 to 16; at week 16, placebo participants were switched to apremilast 30 mg tablets BID for 36 weeks (from week 16 to week 52)
  Interventions: Drug: Placebo; Drug: Placebo-Apremilast

INTERVENTIONS:
Drug: Apremilast — Apremilast 30 mg tablets orally twice daily (BID) weeks 0 to 52.
  Other Names: CC-10004, Otzela
  Arms: Apremilast
Drug: Placebo — Participants randomized to the placebo treatment group received placebo tablets (identical in appearance to the apremilast 30 mg tablets) orally BID for from weeks 0-16.
Drug: Placebo-Apremilast — At Week 16, those randomized to placebo were switched to apremilast 30mg BID for an additional 36 weeks (52 weeks total)
  Other Names: Otezla; CC-10004

SUMMARY:
This study will evaluate the clinical efficacy, the patients quality of life, and safety of oral apremilast 30 mg twice daily (BID) compared to placebo, in adult patients with moderate plaque psoriasis during the 16 week Placebo controlled Phase and then upto 1 year in the Extension Phase of the trial.

DETAILED DESCRIPTION:
This is a Phase 4, multicenter, randomized, placebo-controlled, double-blind study of the efficacy and safety of apremilast in subjects with moderate plaque psoriasis. 221 participants were randomized 2 (apremilast):1 (placebo) at approximately 25 sites in the United States. Those randomized to the apremilast treatment group received apremilast 30 mg tablets orally twice daily for 52 weeks. Those randomized to the placebo treatment group received placebo tablets (identical in appearance to the apremilast 30 mg tablets) orally twice daily (BID) for 16 weeks. Beginning Week 16, those initially randomized to placebo were switched to receive apremilast 30 mg BID for an additional 36 weeks (52 weeks total).

Study enrolled adult patients with stable moderate plaque psoriasis, who are naïve to systemic psoriasis treatments.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females, ≥ 18 years of age at the time of signing the informed consent document.
2. Understand and voluntarily sign an informed consent document prior to any study related assessments/procedures being conducted.
3. Able to adhere to the study visit schedule and other protocol requirements.
4. Diagnosis of chronic plaque psoriasis for at least 6 months prior to signing the informed consent.
5. Have moderate plaque psoriasis at screening and baseline as defined by

   1. BSA (Body Surface Area)5% to 10% and
   2. sPGA (Physician's Global Assessment) 3 (moderate) based on a 0 to 5 point scale
6. Must be in general good health (except for psoriasis) as judged by the investigator, based on medical history, physical examination, and clinical laboratories.
7. No prior exposure to systemic treatments or biologics for the treatment of psoriatic arthritis, psoriasis, or any other indication that could impact the assessment of psoriasis.
8. Females of childbearing potential (FCBP)must have a negative pregnancy test at Screening and Baseline. While on investigational product and for at least 28 days after taking the last dose of investigational product, FCBP who engage in activity in which conception is possible must use one of the approved contraceptive§ options described below: Option 1: Any one of the following highly effective methods: hormonal contraception (oral, injection, implant, transdermal patch, vaginal ring); intrauterine device (IUD); tubal ligation; or partner's vasectomy; OR Option 2: Male or female condom (latex condom or nonlatex condom NOT made out of natural [animal] membrane [for example, polyurethane]) PLUS one additional barrier method: (a) diaphragm with spermicide; (b) cervical cap with spermicide; or (c) contraceptive sponge with spermicide.
9. Male subjects (including those who have had a vasectomy) who engage in activity in which conception is possible must use barrier contraception (male latex condom or nonlatex condom NOT made out of natural [animal] membrane [for example, polyurethane]) while on investigational product and for at least 28 days after the last dose of investigational product

Exclusion Criteria:

1. Other than psoriasis, any clinically significant (as determined by the Investigator) cardiac, endocrinologic, pulmonary, neurologic, psychiatric, hepatic, renal, hematologic,immunologic disease, or other major disease that is currently uncontrolled.
2. Any condition, including the presence of laboratory abnormalities, which would place the subject at unacceptable risk if he/she were to participate in the study.
3. Any condition, including other inflammatory diseases or dermatologic conditions, which confounds the ability to interpret data from the study, including other types of psoriasis (ie, erythrodermic, guttate, inverse, or pustular psoriasis), other than plaque psoriasis.
4. Prior history of suicide attempt at any time in the subject's life time prior to signing the informed consent and randomization, or major psychiatric illness requiring hospitalization within the last 3 years prior to signing the informed consent.
5. Pregnant or breast feeding.
6. Active substance abuse or a history of substance abuse within 6 months prior to signing the informed consent.
7. Malignancy or history of malignancy, except for:

   1. treated (ie, cured) basal cell or squamous cell in situ skin carcinomas;
   2. treated (ie, cured) cervical intraepithelial neoplasia (CIN) or carcinoma in situ of the cervix with no evidence of recurrence within 5 years of signing the informed consent.
8. Topical therapy within 2 weeks of randomization (including, but not limited to, topical corticosteroids, retinoids or vitamin D analog preparations, tacrolimus, pimecrolimus, or anthralin/dithranol). Use of phototherapy within 4 weeks prior to randomization.
9. Use of any investigational drug within 4 weeks prior to randomization, or 5 pharmacokinetic/pharmacodynamic half-lives, if known (whichever is longer).
10. Prolonged sun exposure or use of tanning booths, which may confound the ability to interpret data from the study.
11. Prior treatment with apremilast.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 221 (Actual)
Dates: Start 2015-04-20 (Actual); Primary Completion 2016-02-12 (Actual); Study Completion 2016-11-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (26):
- United States (26):
  - UAB at Birmingham - The Kirklin Clinic, Birmingham, Alabama
  - Center For Dermatology, Fremont, California
  - Dermatology Research Associates, Los Angeles, California
  - Blue Harbor Dermatology, Newport Beach, California
  - Center for Dermatology and Laser Surgery, Sacramento, California
  - East Bay Rheumatology Medical, San Leandro, California
  - Tien Q. Nguyen MD Inc, Tustin, California
  - UConn Health Center, Farmington, Connecticut
  - Dermatology Associates, Panama City, Florida
  - USF Health Faculty Office Building-FOB, Tampa, Florida
  - Forward Clinical Trials Inc, Tampa, Florida
  - Dermatologic Surgery Specialists, P.C., Macon, Georgia
  - Shideler Clinical Research Center, Carmel, Indiana
  - Dermatology Specialists, PSC, Louisville, Kentucky
  - DermResearch, PLLC, Louisville, Kentucky
  - Lawrence Green, MD, LLC, Rockville, Maryland
  - Henry Ford Hospital, Detroit, Michigan
  - Las Vegas Skin and Cancer Clinics, Las Vegas, Nevada
  - Psoriasis Treatment Center of Central New Jersey, East Windsor, New Jersey
  - Garden City Dermatology, Garden City, New York
  - Sadick Research Group, New York, New York
  - Dermatology Associates of Rochester PC, Rochester, New York
  - University of Cincinnati, Cincinnati, Ohio
  - Dermatology and Laser Center of Charleston, Charleston, South Carolina
  - University of Utah School of Medicine, Salt Lake City, Utah
  - Dermatology Consultants, Inc., Lynchburg, Virginia

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- [Background] Reich K, Mrowietz U, Menter A, Griffiths CEM, Bagel J, Strober B, Nunez Gomez N, Shi R, Guerette B, Lebwohl M. Effect of baseline disease severity on achievement of treatment target with apremilast: results from a pooled analysis. J Eur Acad Dermatol Venereol. 2021 Dec;35(12):2409-2414. doi: 10.1111/jdv.17520. Epub 2021 Aug 23. PMID 34255891
- [Derived] Mease PJ, Hatemi G, Paris M, Cheng S, Maes P, Zhang W, Shi R, Flower A, Picard H, Stein Gold L. Apremilast Long-Term Safety Up to 5 Years from 15 Pooled Randomized, Placebo-Controlled Studies of Psoriasis, Psoriatic Arthritis, and Behcet's Syndrome. Am J Clin Dermatol. 2023 Sep;24(5):809-820. doi: 10.1007/s40257-023-00783-7. Epub 2023 Jun 14. PMID 37316690
- [Derived] Stein Gold L, Bagel J, Lebwohl M, Jackson JM, Chen R, Goncalves J, Levi E, Duffin KC. Efficacy and Safety of Apremilast in Systemic- and Biologic-Naive Patients With Moderate Plaque Psoriasis: 52-Week Results of UNVEIL. J Drugs Dermatol. 2018 Feb 1;17(2):221-228. PMID 29462231

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants enrolled into this study were those with moderate plaque psoriasis without prior treatment with systemic agents or biologics and were enrolled across 25 study centers in the United States.
Pre-assignment Details: Participants were randomized in a 2 to 1 ratio to receive apremilast or placebo.
Groups:
- Apremilast: Participants were initially randomized to apremilast (APR) 30 mg tablets twice daily (BID) during the placebo-controlled phase (Weeks 0-16).
- Placebo: Participants were initially randomized to identically matching placebo (PBO) tablets twice a day (BID) during the placebo-controlled phase (Weeks 0-16)
- Placebo-Apremilast: Participants who were initially randomized to receive placebo were switched to apremilast 30 mg PO BID beginning at Week 16, for an additional 36 weeks (52 weeks total).
Period: Placebo-controlled Phase (Week 0 - 16)
Arm/Group | Apremilast | Placebo | Placebo-Apremilast
Started | 148 | 73 | 0
Intent to Treat | 147 (ITT = includes participants who received at least one dose of study drug.) | 73 (ITT = includes participants who received at least one dose of study drug.) | 0
Completed | 121 (Completed = participants who completed Week 16) | 64 (Completed = participants who completed Week 16) | 0
Not Completed | 27 | 9 | 0
Not completed — Adverse Event | 5 | 2 | 0
Not completed — Lack of Efficacy | 0 | 1 | 0
Not completed — Withdrawal by Subject | 9 | 1 | 0
Not completed — Lost to Follow-up | 10 | 4 | 0
Not completed — Other | 3 | 1 | 0
Period: Apremilast Extension Phase (Weeks 16-52)
Arm/Group | Apremilast | Placebo | Placebo-Apremilast
Started | 121 | 0 | 64
Received Treatment | 121 | 0 | 64
Completed | 86 | 0 | 50
Not Completed | 35 | 0 | 14
Not completed — Adverse Event | 7 | 0 | 2
Not completed — Lost to Follow-up | 8 | 0 | 6
Not completed — Withdrawal by Subject | 12 | 0 | 4
Not completed — Lack of Efficacy | 8 | 0 | 1
Not completed — miscellaneous | 0 | 0 | 1
Period: Post-Treatment Observational Follow-Up
Arm/Group | Apremilast | Placebo | Placebo-Apremilast
Started | 81 | 0 | 49
Completed | 80 | 0 | 49
Not Completed | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The intent to treat (ITT) population consisted all participants who were randomized. Participants were included in the treatment arm which they were randomized into the ITT population.
Groups:
- Placebo: Participants were initially randomized to identically matching placebo (PBO) tablets BID during the placebo-controlled phase (Weeks 0-16)
- Total: Total of all reporting groups
Arm/Group | Placebo | Apremilast | Total
Number analyzed (Participants) | 73 | 148 | 221
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 60 | 120 | 180
  >=65 years | 13 | 28 | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.1 (13.74) | 48.6 (15.41) | 49.4 (14.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 74 | 106
  Male | 41 | 74 | 115
Body Surface Area (BSA) [Mean (Standard Deviation); unit: percent affected] — Body Surface Area (BSA) is a measurement of involved skin. The overall BSA affected by psoriasis is estimated based on the palm area of the participant's hand (entire palmar surface or "handprint"), which equates to approximately 1% of total body surface area.
  percent affected | 7.1 (1.75) | 7.2 (1.61) | 7.2 (1.66)
Static Physician's Global Assessment (sPGA) Score [Number; unit: Participants] — The Static Physician's Global Assessment (sPGA) is the assessment by the investigator of the overall disease severity at the time of evaluation. The National Psoriasis Foundation Psoriasis Score version of a static PGA is calculated by averaging the total body erythema, induration, and desquamation scores. Erythema (E), induration (I), and desquamation (D) are scored on a 6-point scale, ranging from 0 (clear) to 5 (very severe), with an overall sPGA calculated as (E + I + D)/3. Scores for each assessment are rounded to the nearest whole number to result in the final score.
  Participants
    1 = Almost Clear | 0 | 0 | 0
    2 = Mild | 0 | 0 | 0
    3 = Moderate | 70 | 144 | 214
    4 =Severe | 3 | 3 | 6
    5 = Very Severe | 0 | 0 | 0
    Missing | 0 | 1 | 1
Product of BSA and sPGA [Mean (Standard Deviation); unit: psoriasis severity index] — For each participant, the product of BSA and sPGA were calculated as BSA value multiplied by the sPGA score (BSA*sPGA), measured as the total psoriasis severity index. The ranges for BSA* sPGA scores were from 15 to 40% for the placebo and apremilast arms respectively. Those in the study who had a baseline BSA in the range of 5-10% and a sPGA score of 3 or 4 were enrolled. Those with a higher psoriasis severity index represented worse outcomes. The difference between participants enrolled (148) in the apremilast group and treated (147) lies in one participant, who was randomized in error.
  psoriasis severity index | 21.6 (5.87) | 21.8 (5.17) | 21.7 (5.40)
Duration of Psoriasis [Mean (Standard Deviation); unit: years] — The difference between participants enrolled (148) in the apremilast group and treated (147) lies in one participant, who was randomized in error.
  years | 12.85 (12.350) | 17.02 (14.138) | 15.64 (13.684)
Ethnicity [Number; unit: participants]
  Hispanic or Latino | 4 | 13 | 17
  Not Hispanic or Latino | 69 | 134 | 203
  Unknown | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Mean Percentage Change From Baseline in the Product of BSA (%) and the sPGA Which is Considered as the Total Psoriasis Severity Index at Week 16
Description: BSA is a measurement of involved skin. The overall BSA affected by psoriasis is estimated based on the palm area of the participant's hand (entire palmar surface or "handprint" including the fingers), which equates to approximately 1% of total body surface area. The sPGA is a 6-point scale ranging from 0 (clear), 1 (almost clear), 2 (mild), 3 (moderate), to 4 (severe), 5 (very severe) incorporating a separate assessment of the severity of the three primary signs of the plaques of all involved areas: erythema, scaling and plaque elevation with an overall sPGA calculated as (E + I + D)/3. Scores for each assessment are rounded to the nearest whole number to result in the final score. The range of BSA*sPGA mean percentage change from baseline to week 16 (end of phase) were -100 to 344.4 and -100 to 100 for the placebo and apremilast groups respectively. Higher scores represented worse outcomes.
Time Frame: Baseline to Week 16 (end of phase)
Population: The Intent-to-Treat (ITT) population consisted of all participants who were randomized. Participants with a baseline value and at least one post-baseline value were included. A missing value at Week 16 was imputed by last observation carried forward. (LOCF).
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Placebo | Apremilast
Number analyzed (Participants) | 73 | 147
percentage change | -10.17 (64.043) | -48.07 (43.699)
Statistical Analysis 1: Comparison: Placebo vs Apremilast; Test type: Superiority or Other; p < 0.0001, ANCOVA; Based on 2-way ANCOVA with treatment and site as factors and baseline value as covariate; LS Mean Difference = -39.84, 95% CI 2-sided [-54.39 to -25.30]

2. Secondary Outcome: Mean Change From Baseline in the Dermatology Life Quality Index (DLQI) Total Score at Week 16
Description: DLQI is a simple, compact, and practical questionnaire for use in a dermatology clinical setting to assess limitations related to the impact of skin disease. The instrument contains ten items dealing with the participant's skin. With the exception of Item Number 7, the participant responds on a four-point scale, ranging from "Very Much" (score 3) to "Not at All" or "Not relevant" (score 0). Item Number 7 is a multi-part item, the first part of which ascertains whether the participant's skin prevented them from working or studying (Yes or No, scores 3 or 0 respectively), and if "No," then the participant is asked how much of a problem the skin has been at work or study over the past week, with response alternatives being "A lot," "A little," or "Not at all" (scores 2, 1, or 0 respectively). The DLQI total score is derived by summing all item scores, which has a possible range of 0 to 30, with 30 corresponding to the worst quality of life, and 0 corresponding to the best.
Time Frame: Baseline to Week 16 (end of phase)
Population: The ITT population consisted of all participants who were randomized. Participants with a baseline value and at least one post-baseline value are included. A missing value at Week 16 (end of phase) was imputed by LOCF.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Apremilast
Number analyzed (Participants) | 71 | 144
units on a scale | -2.4 (6.62) | -4.8 (5.80)
Statistical Analysis 1: Comparison: Placebo vs Apremilast; Test type: Superiority or Other; p = 0.0008, ANCOVA; Based on 2-way ANCOVA with treatment and site as factors and baseline value as covariate; LS Mean Difference = -2.5, 95% CI 2-sided [-3.9 to -1.0]

3. Secondary Outcome: Percentage of Participants Who Achieved a sPGA Score of Clear (0) or Almost Clear (1) at Week 16 From Baseline
Description: The sPGA is an assessment by the investigator of the overall disease severity at the time of evaluation. Erythema (E), induration (I), and desquamation (D) are scored on a 6-point scale, ranging from 0 (clear) to 5 (very severe), with an overall sPGA calculated as (E + I + D)/3. Scores for each assessment are averaged and rounded to the nearest whole number to result in the final sPGA score.
Time Frame: Baseline to Week 16 (end of phase)
Population: The ITT population consisted of all participants who were randomized. Participants with and at least one post-baseline value are included. A missing value at Week 16 was imputed by LOCF.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Apremilast
Number analyzed (Participants) | 73 | 148
percentage of participants | 9.6 [4.7 to 18.5] | 30.4 [23.6 to 38.2]
Statistical Analysis 1: Comparison: Placebo vs Apremilast; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — Two-sided p-value is based on the Cochran-Mantel-Haenszel test stratified by sites; Difference = 21.0, 95% CI 2-sided [11.0 to 31.1] — Two-sided 95% confidence intervals (CI) is based on normal approximation

4. Secondary Outcome: Percentage of Participants Who Achieved a Clear (0) or Very Mild (1) on Patient Global Assessment (PtGA) Scale at Week 16 From Baseline
Description: The PtGA response rate is defined as the percentage of participants achieving 0 (clear) or 1 (very mild) on the PtGA scale at Week 16. The PtGA is the assessment by the participant of the overall disease severity at the time of evaluation. The PtGA is a 5-point scale ranging from 0 (clear) to 4 (severe).
Time Frame: Baseline to Week 16 (end of phase)
Population: The ITT population consisted of all participants who were randomized. Participants with at least one post-baseline value are included. A missing value at Week 16 (end of phase) was imputed by LOCF.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Apremilast
Number analyzed (Participants) | 73 | 148
percentage of participants | 20.5 [12.9 to 31.2] | 33.8 [26.7 to 41.7]
Statistical Analysis 1: Comparison: Placebo vs Apremilast; Test type: Superiority or Other; p = 0.0365, Cochran-Mantel-Haenszel; 2-sided p-value is calculated based on Cochran-Mantel-Haenszel test stratified by sites; Difference = 13.7, 95% CI 2-sided [1.7 to 25.7] — Two-sided 95% CI is based on normal approximation

5. Secondary Outcome: Mean Change From Baseline in Pruritus Visual Analog Scale (VAS)
Description: The Pruritus VAS assessment was conducted at the baseline visit and each post-baseline visit. The participant was asked to place a vertical stroke on a 100 mm VAS on which the left-hand boundary (0) represents no itch, and the right-hand boundary (100) represents itch as severe as can be imagined. The distance from the mark to the left-hand boundary will be recorded. The Pruritus VAS score ranges from 0 to 100. Higher scores correspond to more severe symptom.
Time Frame: Baseline to Weeks 1 and 16 (end of phase)
Population: ITT population consisted of all participants who were randomized. Participants with a baseline value and at least one post-baseline value are included. A missing value at Week 16 (end of phase) was imputed by LOCF.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Apremilast
Number analyzed (Participants) | 73 | 148
units on a scale
  Week 1 | -9.6 (21.50) | -13.9 (20.00)
  Week 16 | -10.2 (30.73) | -19.2 (26.09)
Statistical Analysis 1: Comparison: Placebo vs Apremilast; The treatment comparison was only done for Week 16; End of Phase; Test type: Superiority or Other; p = 0.0016, ANCOVA; Based on 2-way ANCOVA with treatment and site as factors and baseline value as covariate; LS Mean Difference = -11.6, 95% CI 2-sided [-18.8 to -4.5]

6. Secondary Outcome: Percentage of Participants With Scalp Psoriasis Who Achieved a Clear (0) or Minimal (1) on Scalp Physician's Global Assessment (ScPGA) Scale at Week 16.
Description: The ScPGA assessed scalp involvement, if present at baseline. The 6-point ScPGA scale includes three dimensions (Plaque Thickening, Scaling, and Erythema) and a global assessment. Scores range from 0 (clear), 1 (minimal), 2 (mild), 3 (moderate), 4 (severe), to 5 (very severe). Analysis of ScPGA was restricted to the participants with scalp involvement at baseline.
Time Frame: Baseline to Week 16 (end of phase)
Population: The ITT population with scalp psoriasis who were randomized. Participants with at least one post-baseline value are included. A missing value at Week 16 (end of phase) was imputed by LOCF.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Apremilast
Number analyzed (Participants) | 55 | 112
percentage of participants | 38.2 [26.5 to 51.4] | 50.0 [40.9 to 59.1]
Statistical Analysis 1: Comparison: Placebo vs Apremilast; Test type: Superiority or Other; p = 0.0463, Cochran-Mantel-Haenszel; p-value was based on 2-sided CMH tests stratified by sites; Difference = 11.8, 95% CI 2-sided [-4.0 to 27.6] — Two-sided 95% CI is based on normal approximation

7. Secondary Outcome: Treatment Satisfaction Questionnaire for Medication (TSQM) Version II at Week 16
Description: The TSQM version II is an 11-question self-administered instrument to understand a participation's satisfaction with the current therapy. The TSQM scale comprises four domains, on which participants evaluate their medication (i.e., effectiveness, side effects, convenience and global satisfaction. TSQM scores range from 0 to 100 for each domain; a higher score mean indicates higher satisfaction with treatment.
Time Frame: Baseline to Week 16 (end of phase)
Population: The ITT population consisted of all participants who were randomized. Participants with at least one post-baseline value are included. A missing value at Week 16 (end of phase) was imputed LOCF.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Apremilast
Number analyzed (Participants) | 73 | 146
units on a scale
  TSQM-Effectiveness | 38.81 (25.843) | 57.25 (26.484)
  TSQM-Side Effects | 75.00 (32.428) | 78.50 (20.858)
  TSQM-Convenience | 65.68 (16.650) | 66.93 (21.216)
  TSQM-Global Satisfaction | 48.74 (25.673) | 63.24 (23.624)
Statistical Analysis 1: Comparison: Placebo vs Apremilast; TSQM-Effectiveness; Test type: Superiority or Other; p < 0.0001, ANOVA; Based on 2-way ANOVA with treatment and site as factors; LS Mean Difference = 17.80, 95% CI 2-sided [10.36 to 25.24]
Statistical Analysis 2: Comparison: Placebo vs Apremilast; TSQM - Side Effects; Test type: Superiority or Other; p = 0.3433, ANOVA; Based on 2-way ANOVA with treatment and site as factors; LS Mean Difference = 5.00, 95% CI 2-sided [-5.40 to 15.40]
Statistical Analysis 3: Comparison: Placebo vs Apremilast; TSMQ-Convenience; Test type: Superiority or Other; p = 0.6250, ANOVA; Based on 2-way ANOVA with treatment and site as factors; LS Mean Difference = 1.40, 95% CI 2-sided [-4.25 to 7.06]
Statistical Analysis 4: Comparison: Placebo vs Apremilast; TSQM-Global Satisfaction; Test type: Superiority or Other; p < 0.0001, ANOVA; Mean Difference (Final Values) = 14.07, 95% CI 2-sided [7.16 to 20.97]

8. Secondary Outcome: Treatment Satisfaction Questionnaire for Medication (TSQM) Version II at Week 52
Description: The TSQM version II is an 11-question self-administered instrument to understand a participants satisfaction on the current therapy. The TSQM scale comprises four domains, on which participants evaluate their medication (i.e., effectiveness, side effects, convenience and global satisfaction. TSQM scores range from 0 to 100 for each domain; a higher score indicates higher satisfaction with treatment.
Time Frame: Baseline to week 52
Population: Apremilast participants who entered and were treated in the apremilast extension phase.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo-Apremilast | Apremilast
Number analyzed (Participants) | 64 | 121
units on a scale
  TSQM-Effectiveness | 57.68 (26.879) | 54.13 (26.898)
  TSQM-Side Effects | 77.29 (27.541) | 75.45 (24.904)
  TSQM-Convenience | 72.74 (17.222) | 71.76 (19.359)
  TSQM-Global Satisfaction | 59.24 (27.941) | 59.92 (27.053)

9. Secondary Outcome: Mean Percentage Change From Baseline in Psoriasis Area Severity Index Score (PASI) at Week 16
Description: The PASI score is a measure of psoriatic disease severity taking into account qualitative lesion characteristics (erythema, thickness, and scaling) and degree of skin surface area involvement on defined anatomical regions. Erythema, thickness, and scaling are scored on a scale of 0 (none) to 4 (very severe) on 4 anatomic regions of the body: head, trunk, upper limbs, and lower limbs. Degree of involvement on each of the 4 anatomic regions is scored on a scale of 0 (no involvement) to 6 (90% to 100% involvement). PASI scores range from 0 to 72, with higher scores reflecting greater disease severity.
Time Frame: Baseline to Week 16 (end of phase)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Placebo | Apremilast
Number analyzed (Participants) | 73 | 147
percentage change | -3.87 (79.441) | -40.72 (49.523)
Statistical Analysis 1: Comparison: Placebo vs Apremilast; Test type: Superiority or Other; p < 0.0001, ANCOVA; Based on 2-way ANCOVA with treatment and site as factors and baseline value as covariate; LS Mean Difference = -37.0, 95% CI 2-sided [-54.08 to -19.91]

10. Secondary Outcome: Percentage of Participants Who Achieved at Least a 50% Improvement (Response) in the Psoriasis Area and Severity Index (PASI)-50 From Baseline at Week 16.
Description: as for outcome 9
Time Frame: Baseline to Week 16 (end of phase)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Apremilast
Number analyzed (Participants) | 73 | 148
percentage of participants | 24.7 [16.2 to 35.6] | 53.4 [45.4 to 61.2]
Statistical Analysis 1: Comparison: Placebo vs Apremilast; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel; 2-sided p-value is calculated based on Cochran-Mantel-Haenszel test stratified by sites; Difference = 29.1, 95% CI 2-sided [16.3 to 41.8] — Two-sided 95% CI is based on normal approximation

11. Secondary Outcome: Percentage of Participants Who Achieved at Least a 75% Improvement (Response) in the Psoriasis Area and Severity Index (PASI)-75 From Baseline at Week 16
Description: as for outcome 9
Time Frame: Baseline to Week 16 (end of phase)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Apremilast
Number analyzed (Participants) | 73 | 148
percentage of participants | 8.2 [3.8 to 16.8] | 21.6 [15.8 to 28.9]
Statistical Analysis 1: Comparison: Placebo vs Apremilast; Test type: Superiority or Other; p = 0.0136, Cochran-Mantel-Haenszel; 2-sided Cochran-Mantel-Haenszel test stratified by sites; Difference = 13.5, 95% CI 2-sided [4.4 to 22.7] — 2-sided 95% CI is based on normal approximation

12. Secondary Outcome: Mean Percentage Change From Baseline in the Product of BSA (%) x sPGA at Week 52
Description: BSA is a measurement of involved skin. The overall BSA affected by psoriasis is estimated based on the palm area of the participant's hand (entire palmar surface or "handprint" including the fingers), which equates to approximately 1% of total body surface area. The sPGA is a 6-point scale ranging from 0 (clear), 1 (almost clear), 2 (mild), 3 (moderate), to 4 (severe), 5 (very severe) incorporating a separate assessment of the severity of the three primary signs of the plaques of all involved areas: erythema, scaling and plaque elevation with an overall sPGA calculated as (E + I + D)/3. Scores for each assessment are rounded to the nearest whole number to result in the final score.
Time Frame: Baseline to Week 52
Population: Apremilast participants who entered and were treated in the apremilast extension phase.
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Placebo-Apremilast | Apremilast
Number analyzed (Participants) | 64 | 121
percentage change | -42.23 (93.211) | -55.45 (44.619)

13. Secondary Outcome: Percentage of Participants With Scalp Psoriasis Who Were Initially Randomized to Apremilast and Maintained the Scalp Physician's Global Assessment (ScPGA) Response From Week 16 to Week 52.
Description: The ScPGA will assess scalp involvement, if present at baseline. The 6-point ScPGA scale includes three dimensions (Plaque Thickening, Scaling, and Erythema) and a global assessment with scores range from 0 (clear), 1 (minimal), 2 (mild), 3 (moderate), 4 (severe), to 5 (very severe). Analysis of ScPGA is restricted to the participants with scalp involvement at baseline.
Time Frame: Week 16 to Week 52
Population: Participants who were initially randomized to apremilast and continued through week 52.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Apremilast
Number analyzed (Participants) | 148
percentage of participants
  Responder status at Week 16 | 50.0 [40.9 to 59.1]
  Responder status maintained at Week 52 | 80.4 [68.2 to 88.7]

14. Secondary Outcome: Number of Participants Who Experienced Treatment-Emergent Adverse Events (TEAEs) During the Placebo Controlled Phase
Description: Treatment-Emergent Adverse Events (TEAEs) are defined as any AEs that begin or worsen on or after the start of study drug through 28 days after the last dose of study drug or study treatment discontinuation date, whichever was later. A serious AE (SAE) is any untoward adverse event that is fatal, life-threatening, results in persistent or significant disability or incapacity, requires or prolongs existing in-patient hospitalization, is a congenital anomaly/birth defect, or is a condition that may jeopardize the patient or may require intervention to prevent one of the outcomes listed above.
Time Frame: From first dose of study drug to Week 16; maximum duration of exposure was 20.1 weeks during placebo controlled phase
Population: The safety population includes all participants who were randomized and received at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | Placebo | Apremilast
Number analyzed (Participants) | 73 | 147
participants
  ≥ At Least 1 TEAE | 35 | 92
  ≥ 1 Drug-related TEAE | 21 | 71
  ≥ At Least 1 Severe TEAE | 1 | 3
  ≥ At Least 1 Serious TEAE | 0 | 3
  ≥ 1 Serious Drug-related TEAE | 0 | 0
  ≥ 1 TEAE leading to drug withdrawal | 3 | 5
  ≥ 1 TEAE Leading to drug interruption | 3 | 9
  Any TEAE leading to death | 0 | 0

15. Secondary Outcome: Number of Participants Who Experienced Treatment-emergent Adverse Events (TEAEs) During the Apremilast-Exposure Phase
Description: as for outcome 14
Time Frame: Date of first dose of apremilast during the placebo controlled phase or date of first dose of apremilast after week 16; overall maximum duration of exposure was 61.5 weeks during apremilast-exposure phase
Population: The safety population includes all participants who were randomized and received at least one dose of study drug; apremilast participants as treated.
Measure: Number; unit: participants
Groups:
- Apremilast: Participants treated with placebo initially, completed Week 16, entered and treated with apremilast during the apremilast open-label extension phase.
Arm/Group | Apremilast
Number analyzed (Participants) | 211
participants
  ≥ At Least 1 TEAE | 142
  ≥ 1 Drug-related TEAE | 98
  ≥ At Least 1 Severe TEAE | 5
  ≥ At Least 1 Serious TEAE | 10
  ≥ 1 Serious Drug-related TEAE | 1
  ≥ 1 TEAE leading to drug withdrawal | 14
  ≥ 1 TEAE Leading to drug interruption | 27
  Any TEAE leading to death | 0

ADVERSE EVENTS:
Time Frame: Adverse events are reported for the 16-week PBO-controlled and the apremilast extension phase and monitored from the date of the first dose of apremilast to 12 January2017; maximum duration of exposure was 61.5 weeks during apremilast-exposure phase.
Description: The difference between participants enrolled (148) in the apremilast group and treated (147) lies in one participant, who was randomized in error.
Groups:
- Placebo-Controlled Phase: Apremilast (Weeks 0-16): Participants were initially randomized to apremilast (APR) 30 mg tablets twice daily (BID) during the placebo-controlled phase (Weeks 0-16).
- Placebo-Controlled Phase: Placebo (Weeks 0-16): Participants initially randomized to identically matching placebo tablets PO BID during the placebo-controlled phase. (Weeks 0-16).
- Extension Phase: APR/APR and Placebo/APR (Weeks 0-52): Includes participants initially randomized to apremilast tablets BID in the placebo controlled phase and continued on apremilast (Apremilast/Apremilast), as well as those who were initially randomized to placebo and switched at week 16 (Placebo/Apremilast) to Apremilast 30 mg tablets BID during weeks 16-52
Arm/Group | Placebo-Controlled Phase: Apremilast (Weeks 0-16) | Placebo-Controlled Phase: Placebo (Weeks 0-16) | Extension Phase: APR/APR and Placebo/APR (Weeks 0-52)
Serious Adverse Events (participants affected / at risk) | 3/147 | 0/73 | 10/211
Other Adverse Events (participants affected / at risk) | 73/147 | 23/73 | 101/211
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo-Controlled Phase: Apremilast (Weeks 0-16) (N=147) | Placebo-Controlled Phase: Placebo (Weeks 0-16) (N=73) | Extension Phase: APR/APR and Placebo/APR (Weeks 0-52) (N=211)
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 1
Pyelonephritis (Infections and infestations) | 1 | 0 | 1
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 1
Suicide attempt (Psychiatric disorders) | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo-Controlled Phase: Apremilast (Weeks 0-16) (N=147) | Placebo-Controlled Phase: Placebo (Weeks 0-16) (N=73) | Extension Phase: APR/APR and Placebo/APR (Weeks 0-52) (N=211)
Diarrhoea (Gastrointestinal disorders) | 43 | 12 | 59
Nausea (Gastrointestinal disorders) | 26 | 7 | 40
Vomiting (Gastrointestinal disorders) | 9 | 2 | 12
Nasopharyngitis (Infections and infestations) | 5 | 2 | 22
Upper respiratory tract infection (Infections and infestations) | 10 | 3 | 15
Decreased appetite (Metabolism and nutrition disorders) | 6 | 4 | 11
Headache (Nervous system disorders) | 30 | 8 | 32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Results from a center cannot be submitted for publication before results of multicenter study are published unless it is more than 1 year since study completion. Then, Investigator can publish if manuscript is submitted to Celgene 60 days prior to submission. If Celgene decides publication would hinder drug development, Investigator must delay submission for up to 90 days. Investigator must delete confidential information before submission or defer publication to permit patent applications.